CLINICAL TRIAL: NCT04305613
Title: Cardiotoxicity in Locally Advanced Lung Cancer Patients Treated With Chemoradiation Therapy: A Prospective Longitudinal Cohort
Brief Title: Cardiotoxicity in Locally Advanced Lung Cancer Patients Treated With Chemoradiation Therapy
Acronym: CLARITY
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 13519
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cardiotoxicity; Lung Cancer Stage III; Lung Cancer Stage II; Radiation Toxicity
Keywords: Radiation Therapy Cardiotoxicity; Cardiovascular Risk Factors; Lung Cancer; Cardiovascular Phenotyping; Radiation Therapy; Cardiovascular Disease; Cardio-Oncology
MeSH Terms: conditions — Cardiotoxicity; Lung Neoplasms; Radiation Injuries; Cardiovascular Diseases | interventions — Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, and Buffy coat will be collected for planned biomarker analysis. Patients may optionally consent to have remaining blood banked for future analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: Patients with locally advanced non-small cell lung cancer
  Interventions: Other: Chemoradiation

INTERVENTIONS:
Other: Chemoradiation — Patients will be treated with definitive concurrent chemoradiation with curative intent as determined by their medical and radiation oncologists. We will consider timing of initiation and discontinuation, type, and cumulative dose of platinum based chemotherapy. We will also consider dose, duration, and type of immunotherapy. Radiation therapy will be delivered via proton or proton therapy. Our primary radiation therapy dose-volume exposures are whole heart volumetric dose. As secondary exposures, we will comprehensively define radiation therapy dose parameters to the right ventricle, entire left ventricle, left ventricle segments, coronary arteries, and mean heart dose.

SUMMARY:
This observational cohort will evaluate the cardiovascular effects of chemoradiation used to treat locally advanced, non-small cell lung cancer. Patients will be enrolled prior to the start of therapy and followed during and for at least 2 years after therapy with echocardiograms, nuclear stress tests, blood sampling, and quality of life surveys.

DETAILED DESCRIPTION:
Lung cancer is both the most common malignancy worldwide and the leading cause of cancer death in the US. While radiation therapy is highly effective for many solid tumors, thoracic radiation therapy carries a risk of cardiovascular morbidity and mortality that limits critical gains in cancer control and survival. The investigators will perform detailed cardiovascular phenotyping using biologic and imaging markers to define functional and physiologic perturbations that occur with radiation therapy. The study will provide insights into how cardiovascular risk factors and disease impact these biologic and functional changes. The investigators will also determine which radiotherapy dose-volume metrics are indicative of subclinical cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically confirmed or clinically diagnosed non-small cell lung cancer where the plan is for definitive treatment that includes radiation
* Able to give written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding
* Prior treatment with anthracyclines
* Radiation treatment not expected to involve any heart exposure as determined by treating provider
* ECOG performance status greater than 2
* Vulnerable patients, including pregnant women and prisoners
* Contraindication to rest/vasodilator stress PET/CT, including: asthma with ongoing wheezing at time of enrollment; known Mobitz Type II AV block, 3rd degree AV block, or sick sinus syndrom, without a pacemaker; systolic blood pressure less than 90mmHg; known hypersensitivity to Regadenoson and adenosine; profound sinus bradycardia (heart rate less than 40bpm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer will be enrolled from the radiation oncology clinics at participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
High Sensitivity C-Reactive Protein | up to 12 months
  Change in hsCRP from baseline
Growth Differentiation Factor 15 | up to 12 months
  Change in GDF-15 from baseline
Placental Growth Factor | up to 12 months
  Change in PIGF from baseline
Left Ventricular Strain | up to 12 months
  Change in echo-derived measures of LV peak systolic strain (longitudinal) from baseline
Ventricular Arterial Coupling | up to 12 months
  Change in echo-derived measures of ventricular-arterial coupling (Ea/Ees) from baseline
Coronary Flow Reserve (CFR_ | 6 months
  Change in PET/CT derived CFR from baseline
Overall Survival (2 Year) | 24 months
  All-cause mortality assessed by electronic medical record (EMR) review
Cardiovascular Specific Mortality (2 Year) | 24 Months
  Cardiovascular specific mortality assessed by EMR review
Major Cardiovascular Events (2 Year) | up to 24 months
  Incidence of MCE assessed by EMR review and patient interview

SECONDARY OUTCOMES:
High-Sensitivity Troponin T | up to 12 months
  Change in hsTnT from baseline
N-type pro Brain Natriuretic Peptide | up to 12 months
  Change in NTproBNP from baseline
Left Ventricular Ejection Fraction (2D) | up to 12 months
  Change in echo-derived LVEF from baseline
Right Ventricular Fractional Area Change (RAC) | up to 12 months
  Change in echo-derived RAC from baseline
Right Ventricular Longitudinal Strain | up to 12 months
  Change in echo-derived RV longitudinal strain from baseline
Circumferential Strain | up to 12 months
  Change in echo-derived circumferential strain from baseline
Diastolic Function | up to 12 months
  Change in echo-derived measures of diastolic function from baseline
Valvular Disease | up to 12 months
  Change in echo-derived measures of valvular disease (degree of regurgitation or stenosis) from baseline
Left Ventricular Ejection Fraction (3D) | up to 12 months
  Change in 3D echocardiography derived LVEF from baseline
Left Ventricular systolic strain (3D) | up to 12 months
  Change in 3D echocardiography derived measures of LV systolic strain from baseline
Left Ventricular Twist and Torsion | up to 12 months
  Change in 3D echocardiography derived measures of LV twist and torsion from baseline
Global and Regional Myocardial Blood Flow at Rest | up to 6 months
  Change in PET/CT derived measures of global and regional myocardial blood flow at rest from baseline
Global and Regional Myocardial Blood Flow at Stress | up to 6 months
  Change in PET/CT derived measures of global and regional myocardial blood flow at stress from baseline
FACIT Fatigue Score | up to 5 years
  Change in FACIT Fatigue score from baseline. Score ranges from 0-52. Higher scores indicated less fatigue.
FACIT Dyspnea Score | up to 5 years
  Change in FACIT Dyspnea score from baseline. Score ranges from 0-30. Higher scores indicate more dyspnea.
Godin Leisure Time Exercise Score | up to 5 years
  Change in Godin Leisure Time Exercise Score from baseline. Higher scores indicate higher levels of physical activity.

OTHER OUTCOMES:
Overall Survival (5 Year) | 5-8 years
  All Cause Mortality assessed by National Death Index Search performed 5 years after the last patient is enrolled.
Cardiovascular Specific Mortality (5 Year) | 5-8 Years
  Cardiovascular Specific Mortality by National Death Index Search performed approximately 5 years after the final patient is enrolled.
Major Cardiovascular Events (5 Year) | 5 years
  Incidence of 5-Year MCE by EMR review and patient interview
NCI Patient Reported Outcomes Common Terms and Criteria for Adverse Events (PRO-CTCAE) | 5 Years
  Incidence of symptomatic adverse events as assessed by NCI's PRO-CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Rutger's University / Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided
Participants may opt in to allowing data and/or banked samples to be used for future research and shared with other researchers. A detailed plan for sharing IPD will be finalized at a later date, and may depend in part on how many participants elect this option. Additional supporting information may be shared, including the study protocol and informed consent form.